CLINICAL TRIAL: NCT06009614
Title: Radicle™ GI Health: A Randomized, Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Gastrointestinal (GI) Health and Other Health Outcomes
Brief Title: Radicle GI Health: A Study of Health and Wellness Products on GI Health and Other Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-2307
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Digestion; Abdominal Pain; GI Disorders
MeSH Terms: conditions — Abdominal Pain; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Placebo Control 1 (Placebo Comparator): GI Health Product Form 1 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 1
- Active Product 1.1 (Experimental): GI Health Product Form 1 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 1.1 Usage
- Placebo Control 2 (Placebo Comparator): GI Health Product Form 2 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 2
- Active Product 2.1 (Experimental): GI Health Product Form 2 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 2.1 Usage
- Active Product 2.2 (Experimental): GI Health Product Form 2 - active product 2
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 2.2 Usage
- Placebo Control 3 (Placebo Comparator): GI Health Product Form 3 - control
  Interventions: Dietary Supplement: Radicle GI Health Placebo Control Form 3
- Active Product 3.1 (Experimental): GI Health Product Form 3 - active product 1
  Interventions: Dietary Supplement: Radicle GI Health Active Study Product 3.1 Usage

INTERVENTIONS:
Dietary Supplement: Radicle GI Health Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Radicle GI Health Active Study Product 1.1 Usage — Participants will use their Radicle GI Health Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Radicle GI Health Placebo Control Form 2 — Participants will use their Radicle GI Health Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Radicle GI Health Active Study Product 2.1 Usage — Participants will use their Radicle GI Health Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Radicle GI Health Active Study Product 2.2 Usage — Participants will use their Radicle GI Health Active Study Product 2.2 as directed for a period of 6 weeks.
  Arms: Active Product 2.2
Dietary Supplement: Radicle GI Health Placebo Control Form 3 — Participants will use their Radicle GI Health Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Radicle GI Health Active Study Product 3.1 Usage — Participants will use their Radicle GI Health Active Study Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1

SUMMARY:
A randomized, blinded, placebo-controlled study assessing the impact of health and wellness products on gastrointestinal (GI) health and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with adult participants, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for less bloating or indigestion, (2) indicate an interest in taking a health and wellness product to potentially help their bloating or indigestion, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data are collected electronically from eligible participants over 7 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, and gender identities
* Resides in the United States
* Endorses less bloating or indigestion as a primary desire
* Has the opportunity for at least 20% improvement in their primary health outcome score
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* The calculated validated health survey (PRO) score during enrollment represents less than mild severity
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports current enrollment in another clinical trial
* Lack of reliable daily access to the internet
* Reports current or recent (within 3 months) use of chemotherapy or immunotherapy
* Reports taking medications with a known moderate or severe interaction with any of the active ingredients studied, or a substantial safety risk: Anticoagulants, antihypertensives, anti-anxiolytics, antidepressants, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs (monoamine oxidase inhibitors), or thyroid products
* Reports a diagnosis of heart disease when a known contraindication exists for any of the active ingredients studied: NYHAA (New York Heart Association) Class III or IV congestive heart failure, Atrial fibrillation, Uncontrolled arrhythmias

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2180 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in GI (Gastrointestinal) - related Quality of Life (QOL) | 6 weeks
  Mean difference in GI-related QOL as assessed by Digestion-associated QOL Questionnaire (DGLQ) (scale 0%-100%; with higher scores corresponding to worse GI-related QOL)

SECONDARY OUTCOMES:
Change in abdominal pain | 6 weeks
  Mean difference in abdominal pain as assessed by Patient Reported Outcome Measurement System (PROMIS) Belly Pain 5A (scale 2-25; with higher scores corresponding to more severe abdominal pain)
Change in gas/bloating | 6 weeks
  Mean Difference in Gas/Bloating as assessed by PROMIS GI Gas and Bloating 13A (scale 2-60; with higher scores corresponding to more severe gas/bloating)
Change in feelings of anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Minimal clinically important difference (MCID) in GI-related QOL | 6 weeks
  Likelihood of experiencing MCID in GI-related QOL as assessed by Digestion-associated QOL Questionnaire (DGLQ)
Minimal clinically important difference (MCID) in abdominal pain | 6 weeks
  Likelihood of experiencing MCID in abdominal pain as assessed by PROMIS Belly Pain 5A
Minimal clinically important difference (MCID) in gas/bloating | 6 weeks
  Likelihood of experiencing MCID in gas/bloating PROMIS GI Gas and Bloating 13A

OTHER OUTCOMES:
Change in mood (emotional distress-depression) | 6 weeks
  Mean difference in emotional distress score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Change in libido | 6 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 2-10; with higher scores corresponding to greater interest in sexual activity)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com